CLINICAL TRIAL: NCT04143009
Title: Adaptation of the Friendship Bench Mental Health Intervention for HIV-infected Perinatal Women in Lilongwe (Periscope)
Brief Title: Adaptation of the Friendship Bench Intervention for HIV-infected Perinatal Women in Lilongwe
Acronym: Periscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Brown University (Other); Ministry of Health, Malawi (Other Government); University of Zimbabwe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-1689; 5R34MH116806-02 (NIH)
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-08

CONDITIONS: Human Immunodeficiency Virus; Perinatal Depression
Keywords: HIV; Depression
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Friendship Bench (EFB) (Experimental): Women seeking ANC services at 2 public health centers in Lilongwe, Malawi will be enrolled into this study arm during study recruitment. Individuals enrolled in this arm will be administered the Enhanced Friendship Bench intervention from date of enrollment through 6 months post-partum.
  Interventions: Behavioral: Enhanced Friendship Bench
- Enhanced Standard Care (ESC) (Active Comparator): Women seeking ANC services at 2 public health centers in Lilongwe, Malawi will be enrolled into this study arm during study recruitment. Individuals enrolled in this arm will received the Enhanced Standard Care intervention from date of enrollment through 6 months post-partum.
  Interventions: Other: Enhanced Standard Care (Control)
- Adapted Friendship Bench (AFB) (Experimental): Women seeking ANC services at 2 public health centers in Lilongwe, Malawi will be enrolled into this study arm during study recruitment. Individuals enrolled in this arm will be administered the Adapted Friendship Bench intervention from date of enrollment through 6 months post-partum.
  Interventions: Behavioral: Adapted Friendship Bench

INTERVENTIONS:
Behavioral: Enhanced Friendship Bench — EFB will include the following: integrating problem solving therapy- based ART adherence support into existing counseling sessions and providing opportunities for participants to address HIV-specific concerns, such as stigma, disclosure, mother-to-child HIV transmission or other issues women identify during counseling sessions, and retention strategies to support engagement in care for HIV-infected women with PND. This intervention will include 4 individual prenatal and 2 group postnatal counseling sessions. To provide additional social support, one support session will be added, at which participants will be invited to bring a person of her choice who can be a support to her in managing both her HIV and/or depression. To assist women with receiving their medication during late pregnancy and postpartum, a trained psychosocial counselor will conduct up to 6 home visits. At each home visit, counselors will be able to deliver a participants' medications and conduct a counseling session.
  Arms: Enhanced Friendship Bench (EFB)
Other: Enhanced Standard Care (Control) — Standard care for mental health in public facilities in Malawi includes options for basic supportive counseling by the primary provider or nurse, medication management by the primary provider, referral to the clinic psychiatric nurse or mental health clinic, or in more severe cases referral to the psychiatric units at tertiary care hospitals. For this study, standard care will be enhanced by a trained study research assistant who will provide mental health evaluation; brief supportive counseling; information, education, and support on common mental disorders; and (if indicated) facilitation of referral to the clinic's psychiatric nurse or mental health clinic. The study research assistant will have up to 3 follow-up contacts with the participant to assess whether she has followed up on recommended referrals or treatment plans and to assess whether any further outreach is indicated.
  Arms: Enhanced Standard Care (ESC)
Behavioral: Adapted Friendship Bench — Adapted Friendship Bench (AFB): AFB will include the following: integrating problem solving therapy- based and antiretroviral therapy (ART) adherence support into existing counseling sessions and providing opportunities for participants to address HIV-specific concerns, such as stigma, disclosure, mother-to-child HIV transmission or other issues women identify during counseling sessions. AFB will include 4 individual prenatal counseling session and 2 group postnatal counseling sessions. No specific retention support will be provided, but participants may identify barriers to engagement in HIV care to address during their pre- or postnatal counseling sessions.
  Arms: Adapted Friendship Bench (AFB)

SUMMARY:
In many sub-Saharan African countries, the scale-up of lifelong antiretroviral treatment (ART) to all pregnant and breastfeeding women under Option B+ has the potential to radically improve maternal health and reduce mother-to-child HIV transmission. However, loss to HIV care after delivery has emerged as an important threat to the hoped-for impact of Option B+. Evidence suggests that one important contributor to postpartum loss to HIV care is perinatal depression (PND). In non-pregnant HIV-infected populations, depression has been linked to poor ART adherence, reduced engagement in care, and ultimately worse HIV clinical outcomes. Thus, interventions that integrate PND treatment with targeted support for HIV care retention are critical to the success of Option B+.

The Friendship Bench is an evidence-based depression counseling intervention delivered by trained, supervised lay health workers. It is proven to reduce depression in the general population in low-resource settings, but has not been adapted to address PND, or enhanced to support engagement in HIV care. The Friendship Bench offers an ideal framework for integrating retention support into a proven depression treatment model. Our long-term goal is to adapt, test, and scale up resource-appropriate interventions to reduce PND and improve engagement in HIV care. The objective of this proposal is to lay the groundwork for an effectiveness trial by adapting the Friendship Bench intervention to address PND and support engagement in care among perinatal HIV-infected women and assessing the feasibility, acceptability, and fidelity of the adapted intervention in Lilongwe, Malawi. In-depth perspectives on PND and its role in engagement in care will be gathered from HIV-infected women with PND, healthcare providers, clinic directors, and Ministry of Health officials using qualitative interviews and focus groups. This formative research will be used to develop an intervention protocol adapted to the unique needs of HIV-infected women during the perinatal period (Adapted Friendship Bench) and further enhanced to support engagement in HIV care (Enhanced Friendship Bench). The Adapted and Enhanced Friendship Bench interventions will be compared to enhanced standard care in a 3-arm pilot study. Feasibility, acceptability, and fidelity will be assessed at 6 months postpartum, along with the interventions' preliminary effectiveness across several mental health and engagement in HIV care measures.

ELIGIBILITY:
Women

Inclusion criteria:

* HIV-infected, pregnant women initiating or re-initiating ART during antenatal care (ANC)
* ≤30 weeks gestation to allow sufficient time for approximately 4 prenatal counseling sessions and approximately 2 postnatal counseling sessions.
* Screened positive for depression with a score > 8 on the Self-Reporting Questionnaire 20-item (SRQ-20)
* At least 18 years of age

Exclusion criteria:

* Women already successfully established on ART will be excluded because they are at a lower risk for disengagement from HIV care.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigators are recruiting pregnant women with perinatal depression
Enrollment: 92 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pence, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- Malawi (3):
  - Mitundu Health Center, Lilongwe, Lilogwe
  - Lumbadzi Health Center, Lilongwe
  - Nathenje Health Center, Lilongwe

IPD SHARING:
Plan to Share IPD: No
The investigators do not intend to share individual participant data (IPD) with other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Adapted Friendship Bench (AFB): 5 women seeking antenatal care (ANC) service at a public health center in Lilongwe, Malawi will be enrolled into this study arm during study recruitment. Individuals enrolled in this arm will be administered the Enhanced Friendship Bench intervention from date of enrollment through 6 months post-partum.
  Adapted Friendship Bench (AFB): AFB will include the following: integrating problem solving therapy- based and antiretroviral therapy (ART) adherence support into existing counseling sessions and providing opportunities for participants to address HIV-specific concerns, such as stigma, disclosure, mother-to-child HIV transmission or other issues women identify during counseling sessions. AFB will include 4 individual prenatal counseling session and 2 group postnatal counseling sessions. No specific retention support will be provided, but participants may identify barriers to engagement in HIV care to address during their pre- or postnatal counseling sessions.
- Enhanced Friendship Bench (EFB): 43 women seeking ANC services at 2 public health centers in Lilongwe, Malawi will be enrolled into this study arm during study recruitment. Individuals enrolled in this arm will be administered the Enhanced Friendship Bench intervention from date of enrollment through 6 months post-partum.
  Enhanced Friendship Bench: EFB will include the following: integrating problem solving therapy- based ART adherence support into existing counseling sessions and providing opportunities for participants to address HIV-specific concerns, such as stigma, disclosure, mother-to-child HIV transmission or other issues women identify during counseling sessions, and retention strategies to support engagement in care for HIV-infected women with perinatal depression (PND). This intervention will include 4 individual prenatal and 2 group postnatal counseling sessions. To provide additional social support, one support session will be added, at which participants will be invited to bring a person of her choice who can be a support to her in managing both her HIV and/or depression. To assist women with receiving their medication during late pregnancy and postpartum, a trained psychosocial counselor will conduct up to 6 home visits. At each home visit, counselors will be able to deliver a participants' medications and conduct a counseling session.
- Enhanced Standard Care (ESC): 44 women seeking ANC services at 2 public health centers in Lilongwe, Malawi will be enrolled into this study arm during study recruitment. Individuals enrolled in this arm will received the Enhanced Standard Care intervention from date of enrollment through 6 months post-partum.
  Enhanced Standard Care [ESC (Control)]: Standard care for mental health in public facilities in Malawi includes options for basic supportive counseling by the primary provider or nurse, medication management by the primary provider, referral to the clinic psychiatric nurse or mental health clinic, or in more severe cases referral to the psychiatric units at tertiary care hospitals. For this study, standard care will be enhanced by a trained study research assistant who will provide mental health evaluation; brief supportive counseling; information, education, and support on common mental disorders; and (if indicated) facilitation of referral to the clinic's psychiatric nurse or mental health clinic. The study research assistant will have up to 3 follow-up contacts with the participant to assess whether she has followed up on recommended referrals or treatment plans and to assess whether any further outreach is indicated.
Period: Pre-pilot
Arm/Group | Adapted Friendship Bench (AFB) | Enhanced Friendship Bench (EFB) | Enhanced Standard Care (ESC)
Started | 5 | 3 | 4
Completed | 5 | 3 | 4
Not Completed | 0 | 0 | 0
Period: Pilot Trial
Arm/Group | Adapted Friendship Bench (AFB) | Enhanced Friendship Bench (EFB) | Enhanced Standard Care (ESC)
Started | 0 (The AFB arm was removed in study period 2 (Pilot trial phase), and thus 0 participants started the trial in the AFB arm.) | 40 (The study protocol was modified to 2 arms with randomization at the individual level. 40 participants started in the EFB arm for study period 2 (Pilot Trial Phase).) | 40 (The study protocol was modified to 2 arms with randomization at the individual level. 40 participants started in the Enhanced Standard Care (ESC) arm for study period 2 (Pilot Trial Phase).)
Completed | 0 | 39 | 39
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Adapted Friendship Bench (AFB): Women seeking ANC service at a public health center in Lilongwe, Malawi will be enrolled into this study arm during study recruitment. Individuals enrolled in this arm will be administered the Enhanced Friendship Bench intervention from date of enrollment through 6 months post-partum.
  Adapted Friendship Bench (AFB): AFB will include the following: integrating problem solving therapy- based ART adherence support into existing counseling sessions and providing opportunities for participants to address HIV-specific concerns, such as stigma, disclosure, mother-to-child HIV transmission or other issues women identify during counseling sessions. AFB will include 4 individual prenatal counseling session and 2 group postnatal counseling sessions. No specific retention support will be provided, but participants may identify barriers to engagement in HIV care to address during their pre- or postnatal counseling sessions.
- Total: Total of all reporting groups
Arm/Group | Adapted Friendship Bench (AFB) | Enhanced Friendship Bench (EFB) | Enhanced Standard Care (ESC) | Total
Number analyzed (Participants) | 5 | 43 | 44 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (6.9) | 29.3 (5.6) | 28.1 (5.9) | 28.3 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 43 | 44 | 92
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 5 | 43 | 44 | 92

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility- Number of Participants Enrolled in Each Arm
Description: This measure of feasibility will be assessed as the number of women enrolled in each arm out of the desired total sample size of 92 women during the 16 month recruitment period.
Time Frame: Study enrollment period of approximately 16 months
Measure: Count of Participants; unit: Participants
Groups:
- Adapted Friendship Bench (AFB): Women seeking ANC service at a public health center in Lilongwe, Malawi will be enrolled into this study arm during study recruitment. Individuals enrolled in this arm will be administered the Enhanced Friendship Bench intervention from date of enrollment through 6 months post-partum.
Arm/Group | Adapted Friendship Bench (AFB) | Enhanced Friendship Bench (EFB) | Enhanced Standard Care (ESC)
Number analyzed (Participants) | 5 | 43 | 44
Participants | 5 | 43 | 44

2. Primary Outcome: Intervention Feasibility- Proportion of Women Retained in Each Study Arm at 6 Months Post-partum
Description: The proportion of enrolled study participants that remain in their assigned study arm at 6-months post-partum.
Time Frame: 6-months post-partum
Measure: Number; unit: proportion of participants
Arm/Group | Adapted Friendship Bench (AFB) | Enhanced Friendship Bench (EFB) | Enhanced Standard Care (ESC)
Number analyzed (Participants) | 5 | 43 | 44
proportion of participants | 1 | 0.98 | 0.98

3. Primary Outcome: Acceptability of Intervention- Proportion of Women Enrolled That Found Intervention Easy to Participate in
Description: The proportion of women in the intervention arm (EFB) that were either "satisfied" or "highly satisfied" with the intervention as reported in the 6-month follow-up survey.
Time Frame: 6 months post-partum
Population: This outcome measures acceptability of the EFB intervention, and as such, acceptability measures were only collected among a subset of EFB participants (n = 15) and does not apply to the AFB or ESC participants.
Measure: Number; unit: proportion of EFB participants
Arm/Group | Adapted Friendship Bench (AFB) | Enhanced Friendship Bench (EFB) | Enhanced Standard Care (ESC)
Number analyzed (Participants) | 0 | 15 | 0
proportion of EFB participants |  | 1 |

4. Primary Outcome: Fidelity to Intervention- Proportion of Observed Intervention Sessions Covering 80% of Intervention Checklist Items
Description: Fidelity will be assessed by members of the Friendship Bench team (DHO or study psychiatrist), by using a checklist of intervention characteristics either during direct monitoring or using audio recording of up to 3 randomly chosen counseling sessions. Scoring either 'meeting expectations' or 'exceeding' expectations' on at least 80% of applicable checklist items during each session will be considered fidelity to the intervention protocol.
Time Frame: Entire study period (Study baseline through 6 months post-partum)
Population: Fidelity to the intervention was assessed at the session level for the EFB arm. Fidelity was not assessed in the AFB arm as this arm was not included in study period 2 (Pilot Trial). Fidelity was not assessed in the ESC arm because the ESC arm did not receive the intervention. A total of 82 out of 208 completed sessions were assessed for fidelity among a randomly selected subset of 27 participants.
Measure: Number; unit: proportion of sessions meeting threshold
Units Other Than Participants: Intervention Sessions
Arm/Group | Adapted Friendship Bench (AFB) | Enhanced Friendship Bench (EFB) | Enhanced Standard Care (ESC)
Number analyzed (Participants) | 0 | 27 | 0
Number analyzed (Intervention Sessions) | 0 | 82 | 0
proportion of sessions meeting threshold |  | 0.83 |

5. Secondary Outcome: Composite Outcome: Proportion of Women Retained in HIV Care With Improved Depression
Description: The investigator will assess a combined outcome at 6 months of whether a woman was retained in HIV care (defined as attending an HIV care appointment within the 30 days prior to the 6-month interview) and had ≥50% improvement in the Self-Reporting Questionnaire-20 (SRQ-20) score from baseline. The SRQ-20 was developed by the World Health Organization and has scores ranging from 0 to 20 and higher scores indicating a greater level of depression. Scores greater than or equal to 8 are typically considered indicative of a common mental disorder (CMD).
  This measure will capture the proportion of enrolled women with the composite outcome of interest described above.
Time Frame: 6 months post-partum
Population: The analysis population for each arm consists of all the participants who completed the 6-month interview. In the AFB arm, 5 of 5 participants completed the interview. In the EFB arm, 42 of 43 participants completed the 6 month interview (1 participant lost to follow up). In the ESC arm, 43 of 44 participants completed the 6 month interview (1 participant lost to follow up).
Measure: Number; unit: proportion of participants
Arm/Group | Adapted Friendship Bench (AFB) | Enhanced Friendship Bench (EFB) | Enhanced Standard Care (ESC)
Number analyzed (Participants) | 5 | 42 | 43
proportion of participants | 0.20 | 0.40 | 0.14

6. Other Pre Specified Outcome: Proportion of Women Reporting a Score Greater Than or Equal to 8 on the Self-Reporting Questionnaire-20 (SRQ-20)
Description: The proportion of women in each arm that score greater than or equal to 8 on the Self-Reporting Questionnaire-20 at a study visit approximately 6-months post-partum. The SRQ-20 was developed by the World Health Organization and has scores ranging from 0 to 20 and higher scores indicating a greater level of depression. Scores greater than or equal to 8 are typically considered indicative of a common mental disorder (CMD).
Time Frame: 6 months post-partum
Population: as for outcome 5
Measure: Number; unit: proportion of participants
Arm/Group | Adapted Friendship Bench (AFB) | Enhanced Friendship Bench (EFB) | Enhanced Standard Care (ESC)
Number analyzed (Participants) | 5 | 42 | 43
proportion of participants | 0.60 | 0.21 | 0.30

7. Other Pre Specified Outcome: Proportion of Women Retained in HIV Care
Description: The proportion of women who attended at least 1 HIV care appointment within 30-days prior to the 6-month interview.
Time Frame: 6 months post-partum
Population: as for outcome 5
Measure: Number; unit: proportion of participants
Arm/Group | Adapted Friendship Bench (AFB) | Enhanced Friendship Bench (EFB) | Enhanced Standard Care (ESC)
Number analyzed (Participants) | 5 | 42 | 43
proportion of participants | 0.20 | 0.50 | 0.26

8. Other Pre Specified Outcome: Proportion of Women Virally Suppressed
Description: The proportion of women in each arm with an HIV viral load of <1,000 copies/mL
Time Frame: 6 months post partum
Population: The analysis population for each arm consists of all the participants who had a viral load sample collected in the 6 month interview study window. In the AFB arm 5/5 participants had a viral load sample collected. In the EFB arm 30/43 women had a viral load sample collected. In the ESC arm, 32/44 women had a sample viral load collected.
Measure: Number; unit: proportion of participants
Arm/Group | Adapted Friendship Bench (AFB) | Enhanced Friendship Bench (EFB) | Enhanced Standard Care (ESC)
Number analyzed (Participants) | 5 | 30 | 32
proportion of participants | 0.8 | 0.93 | 0.91

9. Other Pre Specified Outcome: The Proportion of Women Whose Infants Received an HIV Viral Load Test
Description: The proportion of women in each arm whose infants had received an HIV viral load test by the time of a study visit approximately 6-months post-partum
Time Frame: 6 months post partum
Population: The AFB arm includes 4/5 participants included in the analysis population as there was 1 infant death in the AFB arm.
  The EFB arm includes 38/43 participants included in the analysis population as there were 3 infant deaths, 1 miscarriage, and 1 woman lost to follow up.
  The ESC arm includes 38/44 participants included in the analysis population as there were 2 infant deaths, 2 still births, 1 miscarriage, and 1 woman lost to follow up.
Measure: Number; unit: proportion of participants
Arm/Group | Adapted Friendship Bench (AFB) | Enhanced Friendship Bench (EFB) | Enhanced Standard Care (ESC)
Number analyzed (Participants) | 4 | 38 | 38
proportion of participants | 1 | 0.95 | 0.95

ADVERSE EVENTS:
Time Frame: Adverse events were collected from consent through each participant's study completion, up to approximately 6 months post-delivery.
Arm/Group | Adapted Friendship Bench (AFB) | Enhanced Friendship Bench (EFB) | Enhanced Standard Care (ESC)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/43 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/5 | 4/43 | 5/44
Other Adverse Events (participants affected / at risk) | 0/5 | 0/43 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapted Friendship Bench (AFB) (N=5) | Enhanced Friendship Bench (EFB) (N=43) | Enhanced Standard Care (ESC) (N=44)
Infant Death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3) | 2 (2)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04143009/Prot_SAP_003.pdf
  • Informed Consent Form: Screening (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT04143009/ICF_004.pdf